CLINICAL TRIAL: NCT03794180
Title: First-in-Human, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study of TJ003234 (Anti-Granulocyte-macrophage Colony-stimulating Factor (GM-CSF) Monoclonal Antibody) in Healthy Subjects
Brief Title: Study of TJ003234 (Anti-GM-CSF Monoclonal Antibody) in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: I-Mab Biopharma US Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJ003234RAR101
Record Dates: First submitted 2018-12-28; First posted 2019-01-04 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Healthy Adult Subjects
Keywords: Anti-GM-CSF agents; GM-CSF/GM-CSFR (GM-CSF receptor) antibody; colony-stimulating factor 2; monoclonal antibody
MeSH Terms: interventions — plonmarlimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TJ003234 (Experimental): 0.3 mg/kg, 1 mg/kg, 3 mg/kg, 10 mg/kg via single IV infusion
  Interventions: Drug: TJ003234
- Placebo (Placebo Comparator): 0 mg/kg via single IV infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TJ003234 — Brownish-yellow liquid containing TJ003234, a recombinant humanized immunoglobulin (Ig) G1 monoclonal antibody diluted with normal saline
  Arms: TJ003234
Drug: Placebo — Colorless to slightly brownish-yellow liquid without TJ003234 diluted with normal saline
  Arms: Placebo

SUMMARY:
TJ003234RAR101 is a first-in-human (FIH), single-center, randomized, double-blind, placebo-controlled, single ascending dose study of TJ003234 in healthy adults to determine whether TJ003234 is safe and tolerated when administered as an intravenous (IV) infusion and to determine the maximum dose tolerated (MTD).

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to sign the informed consent form (ICF)
* Healthy subjects 18-70 years of age
* If of childbearing potential, agree to use protocol-specified contraception
* Body mass index (BMI) 19.0-32.0 kg/m^2
* Blood pressure ≤ 139/89 mm Hg
* Subjects are able to follow the study protocol and complete the trial

Exclusion Criteria:

* Current use of tobacco or nicotine-containing products or illicit drug use
* History of severe allergic or anaphylactic reaction to a therapeutic drug or severe seasonal allergies
* Any known pulmonary disease
* Use of any prescription, investigational drugs, herbal supplements, or nonprescription drugs within 1 month or 5 half-lives (whichever is longer) prior to study drug administration, or dietary supplements within 1 week prior to study drug administration, unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study
* Abnormal hematological and chemistry laboratory values >10% above upper limit of normal (ULN) or >10% below the lower limit of normal (LLN). Absolute neutrophil count (ANC) ≤ 1000 cells/mm^3
* Use of any biologic drugs in the last 120 days prior to dosing.
* Immunization with a live or attenuated vaccine within 4 weeks prior to study drug administration
* Prior treatment with any biologic anti-GM-CSF or GM-CSF receptor antagonists
* ADA screening positive
* Subjects who have a history of documented autoimmune disease, even if not clinically severe or never treated with systemic steroids or immunosuppressive agents
* A positive alcohol test and/or urine drug screen for substance of abuse at screening or upon check-in to the clinical site

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Safety Profile: AEs | Up to 85 days after study drug administration
  Incidence of Adverse Events (AEs)
Maximum Tolerated Dose | Up to 85 days after study drug administration
  Determine Maximum Tolerated Dose of TJ003234

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Parameters: Tmax | Up to 85 days after study drug administration
  Time of peak concentration (Tmax)
Pharmacokinetic (PK) Parameters: Cmax | Up to 85 days after study drug administration
  Maximal Concentration (Cmax)
Pharmacokinetic (PK) Parameters: T1/2 | Up to 85 days after study drug administration
  Investigational product (IP) half-life (T1/2)
Pharmacokinetic (PK) Parameters: CL | Up to 85 days after study drug administration
  Investigational Product (IP) Clearance (CL)
Pharmacokinetic (PK) Parameters: AUC∞ | Up to 85 days after study drug administration
  Area under the curve from time zero extrapolated to infinity (AUC∞)
Anti-drug antibodies (ADA) | Up to 85 days after study drug administration
  Incidence and concentration of anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Claire Xu, MD, PhD, Study Director — I-Mab Biopharma
Locations (1):
- Pharmaron, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No